CLINICAL TRIAL: NCT04246008
Title: Effects of Neuromuscular Training on Functional Capacity in Acute Coronary Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, ARGUISUELAS MARTINEZ MARÍA DOLORES, Head of Physiotherapy Department, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEI18/111
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; neuromuscular training; cardiac rehabilitation; functional capacity
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: This is a mixed-design study. It includes a two-group parallel, randomized clinical trial with acute coronary syndrome patients.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular training group (Experimental): This group will receive a 60-min neuromuscular training sessions twice a week, for 10 weeks until the completion of twenty sessions
  Interventions: Other: Neuromuscular training
- Conventional training group (Active Comparator): This group will receive a 60-min convencional cardiac rehabiliation session twice a week, for 10 weeks until the completion of twenty sessions
  Interventions: Other: Conventional strength training

INTERVENTIONS:
Other: Neuromuscular training — The exercise training was developed based on assuring the correct performance of the exercise focusing in motor control.
  Arms: Neuromuscular training group
Other: Conventional strength training — The exercise training was developed based on standard strength training used in cardiac rehabiliation programmes
  Arms: Conventional training group

SUMMARY:
The purpose of this study is to analyse the effects of neuromuscular training on functional capacity in patients with acute coronary syndrome, compared to the classic strength training of the cardiac rehabilitation programs

DETAILED DESCRIPTION:
So far, there are no previous studies that analyze the effects of neuromuscular training on functional capacity in patients with acute coronary syndrome.

Aim: The main objective of this study is to assess the effects of a 10 weeks neuromuscular training vs traditional strength training programme in patients with acute coronary syndrome.

Design: Randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome patients
* Physical activity must have been prescribed

Exclusion Criteria:

* inflammatory cardiac disease
* severe or moderate ventricular dysfunction
* heart failure
* severe arrhytmias
* systemic hypertension >95% percentile
* pulmonary hypertension >40 mmHg
* aortic stenosis
* baseline O2 <90%
* severe valve insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Incremental Shuttle Walking Test | 10 weeks
  Maximum distance reached

SECONDARY OUTCOMES:
Chester Step Test | 10 weeks
  Time performing the test
30 seconds sit-to- stand test | 10 weeks
  Number of repetitions
Changes in hip muscle strength | 10 weeks
  Measured with dynamometer
Cardiopulmonary exercise testing | 10 weeks
  METS achieved in ergometry
Sexual Health Inventory for Men | 10 weeks
  questionnaire score
EQ-5D-5L | 10 weeks
  Health Related Quality of Life measure

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dolores Arguisuelas, Principal Investigator — Cardenal Herrera University
Locations (1):
- Arguisuelas Martinez Maria Dolores, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] EUROASPIRE I and II Group; European Action on Secondary Prevention by Intervention to Reduce Events. Clinical reality of coronary prevention guidelines: a comparison of EUROASPIRE I and II in nine countries. EUROASPIRE I and II Group. European Action on Secondary Prevention by Intervention to Reduce Events. Lancet. 2001 Mar 31;357(9261):995-1001. doi: 10.1016/s0140-6736(00)04235-5. PMID 11293642
- [Background] Skou ST, Roos EM. Good Life with osteoArthritis in Denmark (GLA:D): evidence-based education and supervised neuromuscular exercise delivered by certified physiotherapists nationwide. BMC Musculoskelet Disord. 2017 Feb 7;18(1):72. doi: 10.1186/s12891-017-1439-y. PMID 28173795
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Derived] Valtuena-Gimeno N, Fabregat-Andres O, Martinez-Hurtado I, Martinez-Olmos FJ, Lluesma-Vidal M, Arguisuelas MD, Ferrer-Sargues FJ. A cardiac rehabilitation programme based on neuromuscular training improves the functional capacity of patients with acute coronary syndrome: a preliminary randomised controlled trial. Physiotherapy. 2025 Mar;126:101428. doi: 10.1016/j.physio.2024.101428. Epub 2024 Sep 20. PMID 39549308